CLINICAL TRIAL: NCT02420665
Title: Use of High-Resolution Microendoscopy (HRME) in Patients With Cervical Dysplasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0368; HHSN261200800001E (Other Grant/Funding Number: NCI); 1R01CA186132 (NIH); NCI-2015-00681 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cervical Dysplasia; Abnormal Pap test; Positive human papillomavirus test; HPV; Visual inspection with acetic acid; VIA; Colposcopy; Proflavine; Acetic acid; High-Resolution Microendoscopy; HRME; Phone call
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Proflavine; Colposcopy; Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- High-Resolution Microendoscopy (HRME) + Colposcopy (Experimental): Visual inspection of cervix performed using 3 - 5% acetic acid to the cervix. Participants undergo standard colposcopy and abnormal lesions noted by quadrant. Then 0.01% proflavine applied topically to the cervix. High-resolution microendoscopy (HRME) then performed. HRME images obtained from one visually normal site and from up to 3 visually abnormal lesions based on visual exam and/or colposcopic findings. Study staff follow up with participant by phone one month after procedure.
  Interventions: Drug: Proflavine; Device: HRME Imaging; Behavioral: Phone Call; Procedure: Colposcopy; Drug: Acetic Acid

INTERVENTIONS:
Drug: Proflavine — 0.01% Proflavine applied topically to the cervix after colposcopy and HRME cervical images obtained.
Device: HRME Imaging — HRME images obtained from one visually normal cervical site, and from up to 3 visually abnormal lesions based on exam and/or colposcopic findings.
  Other Names: High-Resolution Microendoscopy
Behavioral: Phone Call — Study staff follow up with participant by phone one month after procedure.
Procedure: Colposcopy — Colposcopy performed after visual inspection of cervix.
Drug: Acetic Acid — 3 - 5% added to cervix before visual inspection.

SUMMARY:
The goal of this clinical research study is to compare a type of imaging called high-resolution microendoscopy (HRME) for detecting abnormal tissue in the cervix to the standard of care, which is visual inspection with acetic acid (VIA) with a colposcopy procedure. Researchers also want to learn if HRME images can show the difference between cancerous tissue and normal cervical tissue.

DETAILED DESCRIPTION:
If you are found to be eligible to take part in this study, you will first have your scheduled VIA and colposcopy. The study doctor will tell you more about this procedure.

You will then have proflavine hemisulfate solution (contrast dye) applied to your cervix. Images will be collected with the probe from the HRME device. The HRME probe is a long thin tube with a camera at the tip. This should add about 10 minutes to the total procedure time.

The HRME images will be stored in an electronic database and used for research. The images will be deidentified and only the MD Anderson staff will have access. This data will be stored in the database indefinitely (forever).

Any abnormal areas found during the VIA and/or colposcopy will be biopsied as part of your standard of care using very small forceps (a medical tool that is like tongs). If the exam shows no abnormalities, a normal area will be biopsied.

The study doctor will talk to you about the results of the HRME imaging, colposcopy, and biopsy/ies.

There will be no change to the planned standard-of-care colposcopy and biopsy.

Researchers will also collect information from your medical record about the colposcopy, surgery, the status of the disease, and demographics (such as your age).

Follow-Up:

About 1 month after the study procedure, the study staff will contact you by phone to ask how you are doing. The call should last about 5 minutes.

Length of Study:

Your active participation in this study will be over after the biopsy.

This is an investigational study. Proflavine hemisulfate is not FDA approved or commercially available. The HRME device is not FDA approved or commercially available. Both are currently being used for research purposes only.

Up to 800 participants will be enrolled in this study. Up to 400 will take part at MD Anderson and up to 400 will take part at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing colposcopy for an abnormal Pap test, positive HPV test or history of cervical dysplasia (CIN or AIS)
2. Women of childbearing potential must have a negative pregnancy test
3. Women who are at least 21 years of age or older
4. Ability to understand and the willingness to provide informed consent and sign a written Informed Consent Document (ICD)

Exclusion Criteria:

1. Women < 21 years of age
2. Women with a known allergy to proflavine or acriflavine
3. Women who are pregnant or nursing
4. Patients unable or unwilling to provide informed consent or sign a written Informed Consent Document (ICD)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Concordance Between the Diagnosis Using HRME Imaging and the Most Severe Histologic Diagnosis ( Concordance rate monitored using method described by Thall et al. (1995)) | 1 day
  To evaluate the performance of HRME imaging compared with existing diagnostic techniques including colposcopy and visual inspection with acetic acid (VIA), a successful outcome is defined as concordance between the diagnosis using HRME imaging and the most severe histologic diagnosis. That is, researchers will calculate the concordance with the participant as the experimental unit rather than the biopsy, as each participant may have more than 1 biopsy. Target concordance rate is 70%. Concordance rate monitored using method described by Thall et al. (1995), and trial stopped if concordance rate is less than 70%.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org